CLINICAL TRIAL: NCT04726176
Title: COVID-19 and Brain Health
Brief Title: COVID-19 and the Brain
Status: Completed | Type: Observational
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Kevin De Pauw, Professor Dr., Vrije Universiteit Brussel
Other Study IDs: 1432020000338
Record Dates: First submitted 2021-01-25; First posted 2021-01-27 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Covid19; Brain; Neurocognition; fMRI
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19: Participants who were admitted to the intensive care unit due to COVID-19 or participants who exhibited "mild" symptoms due to COVID-19 but needed to be hospitalized.
  Interventions: Biological: Exposure to COVID-19
- Healthy control group: Healthy matched participants who never had COVID-19.

INTERVENTIONS:
Biological: Exposure to COVID-19 — To study the exposure of COVID-19 on the brain and executive functioning
  Groups: COVID-19

SUMMARY:
The main objective of this project is:

1. To assess the impact of COVID-19 on the brain and executive functioning.

Twenty adult subjects of UZ Brussels (volunteers), who needed intensive care due to COVID-19 (n=10) or exhibited mild symptoms due to COVID-19 (n=10), will be recruited after hospital discharge. After signing an informed consent the subjects will undergo brain scans (T1, DTI, SWI, DWI, FLAIR MRI and rsfMRI), an emotion regulation task and a neurocognitive test battery. The latter test battery will be performed using an iPad and will test different neurocognitive functions such as memory, abstract thinking, spatial orientation and attention. The duration of the test battery is 18min. The total duration of one trial is estimated at one hour and a half. All tests are planned at the department of Radiology-Magnetic Resonance (UZ Brussel). After three months patients will visit the department of Radiology-Magnetic Resonance a second time for the same experimental trial. Additionally, a matched control group (n = 20; non covid or ICU patients) will be included and undergo the same tests in order to compare the results of the brain scans, emotional regulation task and neurocognitive test battery with results of both Covid-groups. Next to objective data, questionnaires will be filled out, i.e. visual analogue scales of mental and physical fatigue, Profile of Mood States and some additional return to work questions.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of UZ Brussels, who left the hospital and needed intensive care
* Adult patients of UZ Brussels, who left the hospital and exhibited mild symptoms
* Healthy volunteers (who never had COVID-19)
* Ability to give informed consent
* Dutch or French speaking

Exclusion Criteria:

* History of neurological diseases

Ages: 35 Years to 76 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Both the "ICU COVID-19" and "Mild COVID-19" groups will be selected from COVID-19 patients that were admitted to the UZ Brussel hospital.
  The "Healthy volunteers" group will be selected through the network of the involved researchers (convenience sampling).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-01-30 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Brain scans | Up to 12 weeks
  T1, FLAIR MRI, SWI, DWI, DTI, rsfMRI and a task-based functional MRI
Neurocognitive test battery | Up to 12 weeks
  The computerized cognitive test battery "Cognition" will be conducted using an iPad. This cognitive test battery is sensitive to multiple domains at high-level cognitive performance. It consists of the motor praxis test (measure of sensorimotor speed), visual object learning test (measure of spatial learning and memory), abstract matching (measure of abstraction), line orientation test (measure of spatial orientation), digit symbol substitution test (measure of complex scanning and visual tracking), balloon analogue risk test (measure of risk decision making), NBACK (measure of working memory) and psychomotor vigilance test (measure, or vigilant attention) and takes approximately 18 min in total.

SECONDARY OUTCOMES:
Emotion regulation task | Up to 12 weeks
  During the last brain scan, i.e. the task-based functional fMRI, a short emotion regulation task will be employed. Twenty negatively rated stimuli from the International Affective Picture System balanced on arousal (exciting/calm) will be randomly allocated to one of two blocks, one block per condition (experiential awareness, i.e. switching attention towards the bodily felt affective experience / cognitive reappraisal i.e. cognitively changing how one appraises the situation represented on the negative pictures).
Mental fatigue Visual Analogue Scale (M-VAS) | Up to 12 weeks
  Subjective measure of mental fatigue (0-10cm; 0 = no mental fatigue; 10 = maximal mental fatigue)
Physical fatigue Visual Analogue Scale (P-VAS) | Up to 12 weeks
  Subjective measure of physical fatigue (0-10cm; 0 = no mental fatigue; 10 = maximal mental fatigue)
Return to work questionnaire | Up to 12 weeks
  Questionnaire encompassing the following questions:
  1. When did you restart work duties after hospital discharge?
  2. Did you consider yourself fit to return to work?
  3. What is your general experience of restart working?
  4. Have you been equally as productive, less productive, or more productive than before the COVID-19 infection/since the former consultation?
Profile of Mood States (POMS) | Up to 12 weeks
  The Profile of Mood States (POMS) is a 65 item self-report psychological instrument. The POMS measures six different dimensions of mood states over a period of time. These include: Tension or Anxiety, Anger or Hostility, Vigor or Activity, Fatigue or Inertia, Depression or Dejection, Confusion or Bewilderment. These 65 items are rated on a five-point scale ranging from "not at all" to "extremely".

CONTACTS AND LOCATIONS:
Overall Officials: Kevin De Pauw, Prof. Dr., Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- Vrije Universiteit Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Researchers, K De Pauw, R Meeusen, B Tassignon, J De Mey, L Van Liedekerke, H Raeymaekers, F De Ridder, G Nagels, J Van Schependom, M Vandekerckhove, L Van Imschoot, P Lacor, L Seyler, R Mertens, S Allard, AM Van Binst, LCB Fuentes, N Hoornaert, M Naeyaert, A Radwan, P Van Schuerbeek, S Sunaert and E De Waele will have access to IPD.
  All electronic data is stored on the shared encrypted university drive. All files & written data will be stored in a locked filing cabinet. With only the previously mentioned researchers having access.
  All data will be anonymized by assigning an exclusive identity code to each participant. The identity of the individual will only be known by the previously stated research team. Anonymized data will be stored for up to four years to allow for publication access, further analyses and auditing. All personal data, including health questionnaires and signed consent forms, will be destroyed within 12 months of study completion.

REFERENCES:
- [Background] Iadecola C, Anrather J, Kamel H. Effects of COVID-19 on the Nervous System. Cell. 2020 Oct 1;183(1):16-27.e1. doi: 10.1016/j.cell.2020.08.028. Epub 2020 Aug 19. PMID 32882182